CLINICAL TRIAL: NCT06170762
Title: Sodiumhexametaphosphate Versus MTA as Pulp Capping Material for Immature Permanent Teeth ( Randomized Clinical Trial)
Brief Title: Sodiumhexametaphosphate Versus MTA as Pulp Capping Material for Immature Permanent Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mahmoud Ahmed Mahmoud, Lecturer, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 800
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Pulp Disease, Dental
MeSH Terms: conditions — Dental Pulp Diseases | interventions — Dental Pulp Capping; Pemetrexed

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodiumhexametaphosphate (Experimental)
  Interventions: Other: Pulp capping; Drug: Sodiumhexametaphosphate
- MTA (Active Comparator)
  Interventions: Other: Pulp capping; Other: MTA

INTERVENTIONS:
Other: Pulp capping — Pulp capping material for immature permanent teeth in case of carious or traumatic pulp expures
Drug: Sodiumhexametaphosphate — Sodiumhexametaphosphate
  Arms: Sodiumhexametaphosphate
Other: MTA — MTA
  Arms: MTA

SUMMARY:
Sodiumhexametaphosphate will be used as capping material for dental pulp of immature permanent teeth

ELIGIBILITY:
Inclusion Criteria:

* healthy children
* cooperative children
* deep carious lesion
* traumatic pulp exposure
* immature permanent teeth

Exclusion Criteria:

* uncooperative children
* children with systemic disorders
* non vital immature permanent teeth

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2023-12-20 (Estimated); Primary Completion 2024-12-20 (Estimated); Study Completion 2025-01-20 (Estimated)

PRIMARY OUTCOMES:
Clinical success | One year
  Absence of pain, tenderness, mobility and swelling
Radiographic success | One year
  Absence of periapical lesions, internal resorption an external resorption also evidence of continuous root growth